CLINICAL TRIAL: NCT05169437
Title: A Single-Arm Phase-II Study of Niraparib in Locally Advanced or Metastatic Solid Tumor Patients With PALB2 Mutations
Brief Title: Niraparib in the Treatment of Patients With Advanced PALB2 Mutated Tumors
Acronym: PAVO
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Recruitment challenges
Sponsor: Tempus AI (Industry)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TMPS-101; IND Number: 159142 (Other: FDA)
Record Dates: First submitted 2021-12-13; First posted 2021-12-27 (Actual); Results first posted 2025-10-29 (Actual); Last update posted 2025-10-29 (Actual); Status verified 2025-10

CONDITIONS: Solid Tumor; Breast Tumor; Colon Tumor, Malignant; Lung Tumor; Urologic Cancer; Pancreatic Cancer; Melanoma; Metastatic Cancer; Locally Advanced Solid Tumor; Esophageal Cancer; Endometrial Cancer; Head and Neck Cancer
Keywords: PALB2; Solid Tumor; Metastatic Solid Tumor; Locally Advanced Solid Tumor; Advanced Solid Tumor; Local Solid Tumor; PALB2 Mutation; Niraparib; tPALB2; tPALB2 Mutation; Pathogenic tumor; Lung Tumor; Breast Tumor; Colon Tumor; Zejula; Pancreatic Cancer; Urologic Cancer; Melanoma; Metastatic Cancer; Head and Neck Cancer; Endometrial Cancer; Esophageal Cancer
MeSH Terms: conditions — Breast Neoplasms; Colonic Neoplasms; Lung Neoplasms; Urologic Neoplasms; Pancreatic Neoplasms; Melanoma; Neoplasm Metastasis; Esophageal Neoplasms; Endometrial Neoplasms; Head and Neck Neoplasms | interventions — niraparib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Niraparib in Locally Advanced or Metastatic Solid Tumor Patients with PALB2 Mutations (Experimental)
  Interventions: Drug: Niraparib

INTERVENTIONS:
Drug: Niraparib — Eligible participants will receive daily dosing of Niraparib.
  Other Names: Zejula

SUMMARY:
The purpose of this study is to further evaluate the efficacy and safety of niraparib in patients with locally advanced or metastatic solid tumors and a pathogenic or likely pathogenic tumor PALB2 (tPALB2) mutation.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be at least 18 years of age or older.
* Participants must have a histologically or cytologically confirmed diagnosis of locally advanced or metastatic solid tumor(s).
* Participants must have tested positive for a pathogenic or likely pathogenic tPALB2 gene mutation using a CLIA-certified laboratory as described in the Next-Generation Sequencing (NGS) Laboratory Manual.
* Participants who have stable and asymptomatic Central Nervous System (CNS) disease must be receiving a stable (for at least 7 days) or decreasing corticosteroid dose at the time of study entry.
* Participants must submit fresh or archived (collected within 24 months of enrollment) Formalin-Fixed Paraffin-Embedded (FFPE) tumor sample to the central laboratory for post-enrollment confirmation of tPALB2 status.
* Participants must have received all standard therapies appropriate for their tumor type and stage of disease or, in the opinion of the Investigator, the patient would be unlikely to tolerate or derive clinically meaningful benefit from appropriate standard of care therapy, or the participant has no satisfactory alternative treatments.

Exclusion Criteria:

* Participants have other active concomitant malignancy that warrants systemic, biologic, or hormonal therapy.
* Participants who have ovarian or prostate cancer.
* Participants who have variants of undetermined significance (VUS), but not pathogenic variants of PALB2, at the time of screening.
* Participants who relapsed while receiving platinum based therapy in the adjuvant/curative setting.
* Participants progressing within 14-18 weeks while receiving platinum based therapy in the metastatic setting.
* Participants who have received Poly (ADP-ribose) polymerase (PARP) inhibitor(s) in prior lines of treatment.
* Participants with leptomeningeal disease, carcinomatous meningitis, symptomatic brain metastases, or radiologic signs of CNS hemorrhage.
* Participants with germline or somatic BRCA1 or BRCA2 mutations.
* Participant has systolic blood pressure (BP) over 140 mmHg or diastolic BP over 90 mmHg, despite optimal medical therapy.
* Participants have previously or are currently participating in a treatment study of an investigational agent within 3 weeks of the first dose of therapy preceding the study.
* Participants have received prior systemic cytotoxic chemotherapy, biological therapy, or hormonal therapy for cancer, or received radiation therapy within 3 weeks of the first dose therapy preceding the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2022-03-15 (Actual); Primary Completion 2024-08-06 (Actual); Study Completion 2024-08-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Virginia Rhodes, Study Director — Tempus AI, Inc.
Locations (79):
- United States (79):
  - Yuma Regional Medical Center, Yuma, Arizona
  - Highlands Oncology, Springdale, Arkansas
  - Memorial Care Medical Center, Fountain Valley, California
  - St Joseph Heritage Health - Fullerton, Fullerton, California
  - University of California San Diego, La Jolla, California
  - MemorialCare, Long Beach, California
  - Cancer and Blood Specialty Clinic, Los Alamitos, California
  - Cancer and Blood Specialty, Los Alamitos, California
  - University of California Los Angeles, Los Angeles, California
  - St Joseph Health Medical Group - Napa, Napa, California
  - Ventura County Hematology Oncology Specialists, Oxnard, California
  - Sharp Healthcare, San Diego, California
  - Ridley-Tree Cancer Center, Santa Barbara, California
  - St Joseph Health Medical Group - Santa Rosa, Santa Rosa, California
  - Hartford Healthcare, Hartford, Connecticut
  - Eastern Connecticut Hematology and Oncology, Norwich, Connecticut
  - Holy Cross, Fort Lauderdale, Florida
  - Cancer Specialists of North Florida, Jacksonville, Florida
  - Ocala Community Cancer Center, Ocala, Florida
  - University Cancer & Blood Center, Athens, Georgia
  - Hawaii Cancer Care, Honolulu, Hawaii
  - Rush University Medical Center, Chicago, Illinois
  - Northwest Oncology & Hematology, Rolling Meadows, Illinois
  - Fort Wayne Medical Oncology and Hematology, Fort Wayne, Indiana
  - Goshen Health, Goshen, Indiana
  - Community Health Network, Indianapolis, Indiana
  - Beacon Health System, South Bend, Indiana
  - Pontchartrain Cancer Center, Hammond, Louisiana
  - The Center for Cancer and Blood Disorders - Maryland, Bethesda, Maryland
  - Frederick Health, Frederick, Maryland
  - Maryland Oncology Hematology, Rockville, Maryland
  - Southcoast Health, Fairhaven, Massachusetts
  - Sparrow Health, Lansing, Michigan
  - Central Care Cancer Center, Bolivar, Missouri
  - Mosaic Life Care, Saint Joseph, Missouri
  - Oncology Hematology Associates, Springfield, Missouri
  - Nebraska Cancer Specialists, Omaha, Nebraska
  - OptumCare Cancer Care, Las Vegas, Nevada
  - New Jersey Cancer Care and Blood Disorders, Belleville, New Jersey
  - Englewood Health, Englewood, New Jersey
  - Summit Medical Group, Florham Park, New Jersey
  - Novant Health Inc. - Charlotte, Charlotte, North Carolina
  - Southeastern Medical Oncology Center, Goldsboro, North Carolina
  - Novant Health Inc. - Winston-Salem, Winston-Salem, North Carolina
  - Aultman Medical Group, Canton, Ohio
  - TriHealth, Cincinnati, Ohio
  - University Hospitals Seidman, Cleveland, Ohio
  - Cleveland Clinic - Taussig Cancer Center, Cleveland, Ohio
  - OhioHealth, Columbus, Ohio
  - The Toledo Clinic, Toledo, Ohio
  - Oklahoma Cancer Specialists, Tulsa, Oklahoma
  - Oregon Oncology Specialists, Salem, Oregon
  - Gettysburg Cancer Center, Gettysburg, Pennsylvania
  - Bon Secours - St. Francis Cancer Center, Greenville, South Carolina
  - Avera Cancer Institute, Sioux Falls, South Dakota
  - Sanford Health, Sioux Falls, South Dakota
  - Baptist Cancer Center, Memphis, Tennessee
  - Vanderbilt University, Nashville, Tennessee
  - Texas Oncology - Austin Midtown, Austin, Texas
  - Texas Oncology - Austin Central Pharmacy, Austin, Texas
  - Texas Oncology - South Austin, Austin, Texas
  - Mary Crowley Cancer Research, Dallas, Texas
  - Texas Oncology - Baylor Charles A. Sammons Cancer Center, Dallas, Texas
  - The University of Texas Southwestern Medical Center, Dallas, Texas
  - Oncology Consultants, Houston, Texas
  - Texas Oncology - Longview Cancer Center, Longview, Texas
  - Texas Oncology - Palestine Cancer Center, Palestine, Texas
  - Texas Oncology - Paris Cancer Center, Paris, Texas
  - Lumi Research, Sugar Land, Texas
  - Texas Oncology - Tyler Pharmacy, Tyler, Texas
  - Community Cancer Trials of Utah, Ogden, Utah
  - Utah Cancer Specialists, Salt Lake City, Utah
  - Inova Schar Institute, Fairfax, Virginia
  - Hematology Oncology Associates of Fredericksburg, Fredericksburg, Virginia
  - Virginia Cancer Institute, Richmond, Virginia
  - PeaceHealth, Bellingham, Washington
  - Northwest Medical Specialties, Tacoma, Washington
  - ThedaCare, Appleton, Wisconsin
  - SSM Health, Madison, Wisconsin

RESULTS

PARTICIPANT FLOW:
Groups:
- Niraparib in Locally Advanced or Metastatic Solid Tumor Patients with PALB2 Mutations: This was a multicenter single-arm Phase-II study of niraparib in patients with locally advanced or metastatic solid tumors and a confirmed pathogenic or likely pathogenic tumor PALB2 mutation (tPALB2).
Period: Overall Study
Arm/Group | Niraparib in Locally Advanced or Metastatic Solid Tumor Patients with PALB2 Mutations
Started | 22
Completed | 16
Not Completed | 6

BASELINE CHARACTERISTICS:
Arm/Group | Niraparib in Locally Advanced or Metastatic Solid Tumor Patients with PALB2 Mutations
Number analyzed (Participants) | 22
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 6
  >=65 years | 16
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 16
  More than one race | 0
  Unknown or Not Reported | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 21
  Unknown or Not Reported | 0
Baseline Height [Mean (Standard Deviation); unit: cm] | 166.5 (10.31)
Baseline Weight [Mean (Standard Deviation); unit: kg] | 74.46 (19.663)
Baseline ECOG Performance Status [Count of Participants; unit: Participants] — Scoring for baseline Performance Status was performed by the Eastern Cooperative Oncology Group (ECOG) Performance Status Scale, rating 0-5 (ecog-acrin.org/scale). ECOG 0 = Fully active, able to carry on all pre-disease performance without restriction. ECOG 1 = Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work.
  Participants
    ECOG 0 | 7
    ECOG 1 | 15
Cancer Type [Count of Participants; unit: Participants]
  Colon Cancer | 4
  Pancreatic Carcinoma | 4
  Breast Cancer | 3
  Gastric Cancer | 2
  Bile Duct Cancer | 1
  Endometrial Cancer | 1
  Glioma | 1
  Malignant Melanoma | 1
  Neuroendocrine Carcinoma | 1
  Non-Small Cell Lung Cancer | 1
  Renal Cancer | 1
  Sarcoma | 1
  Uterine Cancer | 1
PALB2 Mutation Type [Count of Participants; unit: Participants]
  Germline | 7
  Somatic | 6
  Unknown | 9

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate (ORR) - Independent Central Review (ICR)
Description: To evaluate overall response rate (ORR) as assessed by Independent Central Review (ICR) using RECIST v1.1
Time Frame: Up to 4 years
Population: This endpoint was not assessed due to early study termination. Due to early study termination, data was not submitted for independent central review and therefore the overall response rate was done according to investigator assessment only and no independent central review was performed.
Measure: Count of Participants; unit: Participants
Arm/Group | Niraparib in Locally Advanced or Metastatic Solid Tumor Patients with PALB2 Mutations
Number analyzed (Participants) | 0
Participants | 0

2. Secondary Outcome: Duration of Response (DOR) - Independent Central Review (ICR)
Description: To evaluate duration of response (DOR) as assessed by ICR using RECIST v1.1
Time Frame: Up to 4 years
Population: This endpoint was not assessed due to early study termination. Due to early study termination, data was not submitted for independent central review and therefore the DOR was done according to investigator assessment only and no independent central review was performed.
Measure: Count of Participants; unit: Participants
Arm/Group | Niraparib in Locally Advanced or Metastatic Solid Tumor Patients with PALB2 Mutations
Number analyzed (Participants) | 0
Participants | 0

3. Secondary Outcome: Progression-Free Survival (PFS) - Independent Central Review (ICR)
Description: To evaluate progression-free survival (PFS) as assessed by ICR using Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST v1.1)
Time Frame: Up to 4 years
Population: This endpoint was not assessed due to early study termination. Due to early study termination, data was not submitted for independent central review and therefore the PFS was done according to investigator assessment only and no independent central review was performed.
Measure: Count of Participants; unit: Participants
Arm/Group | Niraparib in Locally Advanced or Metastatic Solid Tumor Patients with PALB2 Mutations
Number analyzed (Participants) | 0
Participants | 0

4. Secondary Outcome: Overall Response Rate (ORR) - Investigator
Description: To evaluate ORR as defined as the proportion of patients who had a partial or complete response (PR or CR) to therapy, as assessed by Investigator using RECIST v1.1 and assessed periodically throughout the treatment period based on imaging every 8 weeks (56 ± 7 days).
Time Frame: 2 years 3 months
Population: This population consisted of all patients (12 out of 22 patients) with measurable disease who received at least 1 dose of study treatment, who had an adequate baseline tumor assessment, and at least 1 follow-up tumor assessment considered evaluable for anti-tumor efficacy using RECIST v1.1 criteria.
Measure: Count of Participants; unit: Participants
Arm/Group | Niraparib in Locally Advanced or Metastatic Solid Tumor Patients with PALB2 Mutations
Number analyzed (Participants) | 12
Participants
  Complete Response (CR) | 0
  Partial Response (PR) | 2
  Stable Disease (SD) | 5
  Progressive Disease (PD) | 5

5. Secondary Outcome: Duration of Response (DOR) - Investigator
Description: To evaluate DOR as assessed by Investigator using RECIST v1.1 defined as from first documentation of objective tumor response (CR or PR) to first documentation of objective tumor progression or death due to any cause.
Time Frame: 2 years 3 months
Population: This population consisted of all patients (2 patients with CR or PR out of the 12 evaluable for response, out of 22 total patients) with measurable disease who received at least 1 dose of study treatment, who had an adequate baseline tumor assessment, and at least 1 follow-up tumor assessment considered evaluable for anti-tumor efficacy using RECIST v1.1 criteria.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Niraparib in Locally Advanced or Metastatic Solid Tumor Patients with PALB2 Mutations
Number analyzed (Participants) | 2
Months | NA [NA to NA] — Due to early study termination, there are a lack of participant events.

6. Secondary Outcome: Progression-Free Survival (PFS) - Investigator
Description: To evaluate PFS as assessed by Investigator using RECIST v1.1 determined from the first dose to the date of first radiographic progression or death from any cause in the absence of progression, whichever occurred first, or were censored.
Time Frame: 2 years 3 months
Population: as for outcome 4
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Niraparib in Locally Advanced or Metastatic Solid Tumor Patients with PALB2 Mutations
Number analyzed (Participants) | 12
Months | 3.3 [1.7 to NA] — Due to early study termination, there are a lack of participant events.

7. Secondary Outcome: Clinical Benefit Rate (CBR) - Investigator and ICR
Description: To evaluate Clinical Benefit Rate (CBR), defined as the percentage of patients who had achieved Complete Response (CR), Partial Response (PR), or Stable Disease (SD) for 8 weeks or more, as assessed by Investigator only (ICR not performed due to early study termination).
Time Frame: 2 years 3 months
Population: Due to early study termination, data was not submitted for independent central review and therefore the CBR was done according to investigator assessment only and no independent central review. This population consisted of all patients (12 out of 22 patients) with measurable disease who received at least 1 dose of study treatment, who had an adequate baseline tumor assessment, and at least 1 follow-up tumor assessment considered evaluable for anti-tumor efficacy using RECIST v1.1 criteria.
Measure: Count of Participants; unit: Participants
Arm/Group | Niraparib in Locally Advanced or Metastatic Solid Tumor Patients with PALB2 Mutations
Number analyzed (Participants) | 12
Participants | 6 [21.1 to 78.9]

8. Secondary Outcome: ORR With Untreated Measurable CNS Lesions - Investigator
Description: To evaluate intracranial ORR in participants with untreated measurable CNS lesions as assessed by Investigator using RECIST v1.1
Time Frame: Up to 4 years
Population: This endpoint was not assessed due to early study termination. Intracranial ORR in patients with untreated measurable CNS was not measured.
Measure: Count of Participants; unit: Participants
Arm/Group | Niraparib in Locally Advanced or Metastatic Solid Tumor Patients with PALB2 Mutations
Number analyzed (Participants) | 0
Participants | 0

9. Secondary Outcome: ORR With Untreated Measurable CNS Lesions - ICR
Description: To evaluate intracranial ORR in participants with untreated measurable CNS lesions as assessed by ICR using RECIST v1.1
Time Frame: Up to 4 years
Population: This endpoint was not assessed due to early study termination. Due to early study termination, data was not submitted for independent central review and therefore the ORR with untreated measurable CNS lesions was not evaluated by independent central review.
Measure: Count of Participants; unit: Participants
Arm/Group | Niraparib in Locally Advanced or Metastatic Solid Tumor Patients with PALB2 Mutations
Number analyzed (Participants) | 0
Participants | 0

10. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events
Description: To evaluate safety and tolerability per the National Cancer Institute Common Terminology Criteria for Adverse Events version 5.0 (NCI-CTCAE v5.0)
Time Frame: 2 years 3 months
Population: The Safety Population consisted of all 22 enrolled patients who took at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Niraparib in Locally Advanced or Metastatic Solid Tumor Patients with PALB2 Mutations
Number analyzed (Participants) | 22
Participants | 22

11. Secondary Outcome: Overall Survival (OS)
Description: To evaluate overall survival (OS) defined as the time from the date of first dose of study drug to the date of death by any cause. Patients who were alive were censored at the date of last contact.
Time Frame: 6 months and 12 months
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: Percentage
Arm/Group | Niraparib in Locally Advanced or Metastatic Solid Tumor Patients with PALB2 Mutations
Number analyzed (Participants) | 12
Percentage
  Overall Survival at 6 Months | 81.8 [44.7 to 95.1]
  Overall Survival at 12 Months | 51.9 [19.8 to 76.7]

ADVERSE EVENTS:
Time Frame: All adverse events (AEs) and serious adverse events (SAEs) were collected and recorded for each patient from the day of signing the main study informed consent form until 30 days after the last dose of study treatment up to 28 months.
Description: Population includes all patients who took at least 1 dose of study drug.
Arm/Group | Niraparib in Locally Advanced or Metastatic Solid Tumor Patients with PALB2 Mutations
All-Cause Mortality (participants affected / at risk) | 1/22
Serious Adverse Events (participants affected / at risk) | 6/22
Other Adverse Events (participants affected / at risk) | 22/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Niraparib in Locally Advanced or Metastatic Solid Tumor Patients with PALB2 Mutations (N=22)
Anaemia (Blood and lymphatic system disorders) | 2
Ascites (Gastrointestinal disorders) | 1
Haematochezia (Gastrointestinal disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
Multiple organ dysfunction syndrome (General disorders) | 1
Sepsis (Infections and infestations) | 1
Acidosis (Metabolism and nutrition disorders) | 1
Seizure (Nervous system disorders) | 1
Hypotension (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Niraparib in Locally Advanced or Metastatic Solid Tumor Patients with PALB2 Mutations (N=22)
Nausea (Gastrointestinal disorders) | 10
Constipation (Gastrointestinal disorders) | 5
Vomiting (Gastrointestinal disorders) | 4
Abdominal pain (Gastrointestinal disorders) | 3
Abdominal pain lower (Gastrointestinal disorders) | 2
Ascites (Gastrointestinal disorders) | 2
Dyspepsia (Gastrointestinal disorders) | 2
Fatigue (General disorders) | 10
Platelet count decreased (Investigations) | 5
Blood creatinine increased (Investigations) | 4
Alanine aminotransferase increased (Investigations) | 3
Blood alkaline phosphatase increased (Investigations) | 3
Aspartate aminotransferase increased (Investigations) | 2
Blood bilirubin increased (Investigations) | 2
Neutrophil count decreased (Investigations) | 2
Weight Decreased (Investigations) | 2
Decreased appetite (Metabolism and nutrition disorders) | 6
Dehydration (Metabolism and nutrition disorders) | 6
Insomnia (Psychiatric disorders) | 8
Anxiety (Psychiatric disorders) | 4
Dizziness (Nervous system disorders) | 5
Headache (Nervous system disorders) | 5
Anaemia (Blood and lymphatic system disorders) | 7
Thrombocytopenia (Blood and lymphatic system disorders) | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 5
Back pain (Musculoskeletal and connective tissue disorders) | 3
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5
Cough (Respiratory, thoracic and mediastinal disorders) | 3
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 2
Hypertension (Vascular disorders) | 5
Tachycardia (Cardiac disorders) | 3
Skin lesion (Skin and subcutaneous tissue disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (3):
  • Study Protocol: Full Study Protocol (2021-12-06): https://cdn.clinicaltrials.gov/large-docs/37/NCT05169437/Prot_000.pdf
  • Study Protocol: Protocol Clarification Letter (2022-07-27): https://cdn.clinicaltrials.gov/large-docs/37/NCT05169437/Prot_001.pdf
  • Statistical Analysis Plan (2023-12-11): https://cdn.clinicaltrials.gov/large-docs/37/NCT05169437/SAP_002.pdf